CLINICAL TRIAL: NCT00381667
Title: A Randomised, Double-blind, Placebo-controlled, Dose Ascending, Five-way Crossover Study, to Examine Efficacy, Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of a Single Administration of Three Inhaled Doses (25, 100 and 400 Âµg) of GW642444M
Brief Title: Study to Assess GW642444 in Asthma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B2C104604
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: safety; GW642444M; Single Dose; pharmacodynamics; pharmacokinetics; GW642444H; tolerability
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- GW642444M 12.5 (Experimental)
  Interventions: Drug: GW642444M
- GW642444M 100mcg (Experimental)
  Interventions: Drug: GW642444M
- GW642444M 400mcg (Experimental)
  Interventions: Drug: GW642444M
- GW642444H 100mcg (Experimental)
  Interventions: Drug: GW642444H
- Placebo (Experimental)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: GW642444M — M salt
  Other Names: GW642444
  Arms: GW642444M 100mcg; GW642444M 12.5; GW642444M 400mcg
Drug: GW642444H — H salt
  Arms: GW642444H 100mcg
Other: placebo — placebo
  Arms: Placebo

SUMMARY:
This is a study of GW642444M, a long-acting beta 2 specific agonist. This study will examine GW642444M via the inhaled route and will assess the efficacy, safety, tolerability, pharmacodynamics and pharmacokinetics of a single administration of three inhaled doses (25, 100 and 400 µg) of GW642444M in persistent asthmatics. This study will be a single-centre, placebo-controlled, dose-ascending, five-way crossover in 30 asthmatic patients.

Key assessments: efficacy, safety, tolerability, pharmacokinetics and pharmacodynamics will be assessed by measurement of FEV1, blood pressure, pulse rate, 12-lead ECGs, clinical laboratory safety tests, collection of adverse events and blood samples.

ELIGIBILITY:
Inclusion criteria:

* Subjects with a documented history of persistent asthma, with the exclusion of other significant pulmonary diseases
* Female subjects of non-child bearing potential (i.e. post-menopausal or surgically sterile)
* Subjects who are current non-smokers, who have not used any inhaled tobacco products (snuff is permitted) in the 12 month period preceding the screening visit and who have a pack history of less than 10 pack years.
* Subjects with clinically stable persistent asthma within the 4 weeks preceding the screening visit and with a screening pre-bronchodilator FEV1 between 60 and 90% predicted (having abstained from bronchodilators for the required period). Predicted values are based on the ECCS 1993 normal ranges
* During the screening visit, subjects must demonstrate the presence of reversible airway disease, defined as an increase in FEV1 of greater than 12.0% over baseline and an absolute change of greater than 300 mL within 30 minutes following a single 400 mcg salbutamol dose.
* Subjects who are currently taking ICS at a total daily dose of 200 to 500 mcg of FP or equivalent ICS

Exclusion criteria:

* Subjects who have a past or present disease, which as judged by the Investigator and the Medical Monitor, which may affect the safety of the subject or outcome of this study
* A screening Holter ECG tracing that reveals clinically concerning arrhythmias (including, but not limited to, ventricular ectopic runs of 4 beats, R on T phenomena, bigeminy, trigeminy).
* A mean QTc(B) value at screening >430 msec (male) / >450 msec (female) or an ECG that is not suitable for QT measurements (e.g. poorly defined termination of the T wave).
* Any adverse reaction including immediate or delayed hypersensitivity to any ß2 agonist or sympathomimetic drug, or known or suspected sensitivity to the constituents of GW642444 inhalation powder (e.g., lactose or COA).
* Subjects weighing < 50 kg
* Subjects who have participated in any GSK study involving administration of COA.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-08; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Adverse events | throughout study
Laboratory safety tests | throughout study
Holter monitoring | throughout study
Vital signs and 12-lead ECG) | throughout study
Mean change from baseline FEV1 24 hours after dosing. | Day 1, on 5 separate occasions
Supine systolic and diastolic blood pressure and supine heart rate | Day 1 on 5 separate occasions
QTc(B)and QTc(F) | Day 1 on 5 separate occasions

SECONDARY OUTCOMES:
Potassium Max decrease from baseline | Day 1 on 5 separate occasions
Mean change from baseline(0-4h)potassium. | Day 1 on 5 separate occasions
Glucose Max increase from baseline | Day 1 on 5 separate occasions
Weighted mean change from baseline (0-4h)glucose | Day 1 on 5 separate occasions
Derived PK parameters: Cmax, Tmax, AUC(0-t), AUC(0-inf),PEFR | Day 1 on 5 separate occasions

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Clayton, Victoria, Australia
- GSK Investigational Site, Wellington, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: B2C104604 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: B2C104604 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: B2C104604 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: B2C104604 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: B2C104604 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: B2C104604 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: B2C104604 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register